CLINICAL TRIAL: NCT02346123
Title: Determination of Genetic Polymorphisms in Chronic Chagas Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Hospital Sao Rafael (Other)
Responsible Party: Principal Investigator, Milena Botelho Pereira Soares, PhD, Hospital Sao Rafael
Other Study IDs: CEP-41-11
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Chagas Disease
Keywords: Chagas disease; Polymorphisms; Biomarkers
MeSH Terms: conditions — Chagas Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, Serum, Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: Group which contains all the patients of the study.
  Interventions: Genetic: Gathering of samples of genetic material

INTERVENTIONS:
Genetic: Gathering of samples of genetic material — The samples will be obtained from peripheral blood mononuclear cells and the genotyping of the polymorphisms will be done by real time PCR.

SUMMARY:
The purpose of this study is to analyze the influence of polymorphisms of the genes CLDN-1 (Claudina-1), LGALS3 (Lectin galactoside-binding soluble 3), SOCS3 (Suppressor of cytokine signaling 3), IL-28B (interleukin-28B), CCL5 (Chemokine C-C ligand 5) in the determination of clinical forms and in the percentage of cardiac fibrosis in patients with Chagas disease.

DETAILED DESCRIPTION:
The Chagas disease, in its chronic phase, can lead to the development of cardiac arrhythmias and dilated cardiomyopathy, which can evolve to heart failure, causing great morbidity and reduction on patient's quality of life. Some patients stay asymptomatic while others develop the cardiac form of the disease (chronic chagasic cardiomyopathy), or other forms, like the digestive (megacolon and megaesophagus) and the mixed form (cardiac and digestive).

The objective of this study is to analyze the association between single nucleotide polymorphisms with the clinical forms and the amount of cardiac fibrosis in patients with Chagas disease.

The polymorphisms will be analyzed by real time PCR (Polymerase Chain Reaction). The genes whose polymorphisms will be analyzed are: galectin-3, SOCS-3, IL-28B, CLDN-1 and CCL5.

The patients shall be accompanied in the specialized outpatient clinics for Chagas disease - Center of Biotechnology and Cell Therapy. They will be submitted to collection of blood samples for biochemical analysis and cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

* Chagas disease diagnosis confirmed by 2 different serologies
* Diagnosis of Chagas disease in both forms: indeterminate and cardiac ones, with and without ventricular dysfunction

Exclusion Criteria:

* Significant aortic stenosis
* Mitral stenosis with a valve area inferior than 1,5 cm2
* Superior or moderated aortic and/or mitral regurgitation
* Chronic use of immunosuppressive agents
* Dialysis treatment of terminal renal failure
* Fever on the last 48 hours or evidence of systemic infection in activity
* Current abusive use of alcohol or illicit drugs
* Any other comorbidities that impact patient's survival within the next 2 years
* Liver disease in activity
* Continuous use of steroids as treatment for chronic obstructive pulmonary disease
* Hematologic, neoplastic or bone diseases
* Homeostasis disturbances
* Inflammatory diseases or chronic infectious diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Presence of polymorphisms of the genes CLDN-1, LGALS3, SOCS3, IL-28B, CCL5 in the different forms of Chagas disease | The outcome measure will be assessed within one month of follow up.
  We will evaluate the presence of polymorphisms of the genes CLDN-1, LGALS3, SOCS3, IL-28B, CCL5 in the different forms of Chagas disease.

SECONDARY OUTCOMES:
Presence of polymorphisms of the genes CLDN-1, LGALS3, SOCS3, IL-28B, CCL5 in subjects with and without myocardial fibrosis | The outcome measure will be assessed within one month of follow up.
  We will evaluate the presence of polymorphisms of the genes CLDN-1, LGALS3, SOCS3, IL-28B, CCL5 in subjects with and without myocardial fibrosis assessed by magnetic resonance.

CONTACTS AND LOCATIONS:
Overall Officials: Milena BP Soares, PhD, Principal Investigator — Hospital São Rafael; Ricardo R dos Santos, PhD, Study Director — Hospital São Rafael; Bruno SF Souza, MD, Msc, Study Chair — Hospital São Rafael; Gabriela S Cruz, Msc, Study Chair — Hospital São Rafael; Ticiana F Larocca, MD, Msc, Study Chair — Hospital São Rafael; Márcia MN Rabelo, MD, Msc, Study Chair — Hospital São Rafael; Luís CL Correia, MD, PhD, Study Chair — Hospital São Rafael
Locations (1):
- Hospital São Rafael, Salvador, Estado de Bahia, Brazil